CLINICAL TRIAL: NCT02807480
Title: Approach-Avoidance Conflict-a Multi-level Predictor for Therapy Response
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laureate Institute for Brain Research, Inc. (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2015-006-02; 1K23MH108707-01A1 (NIH)
Record Dates: First submitted 2016-06-16; First posted 2016-06-21 (Estimated); Results first posted 2024-03-26 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2024-02

CONDITIONS: Generalized Anxiety Disorder
MeSH Terms: conditions — Generalized Anxiety Disorder | interventions — Surveys and Questionnaires; Interviews as Topic; Magnetic Resonance Imaging; Electroencephalography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Exposure-based therapy (Experimental): Participants will complete 10, 90-minute sessions of Exposure-based therapy, conducted using a group format. Each group will include 8-12 participants. Exposure-based therapy seeks to increase abilities to manage anxiety through repeated practice in facing the situations or thoughts that are the focus of worry or fear. All participants will complete computer-based behavioral assessments, surveys and interviews, functional magnetic resonance imaging (fMRI), and electroencephalography (EEG).
  Interventions: Behavioral: Exposure-based therapy; Behavioral: Computer-based behavioral assessment; Behavioral: Surveys and Interviews; Device: Magnetic resonance imaging (MRI); Device: Electroencephalography (EEG)
- Behavioral Activation therapy (Experimental): Participants will complete 10, 90-minute sessions of Behavioral Activation therapy, conducted using a group format. Each group will include 8-12 participants. Behavioral Activation therapy seeks to target behaviors that might maintain or worsen negative mood. All participants will complete computer-based behavioral assessments, surveys and interviews, functional magnetic resonance imaging (fMRI), and electroencephalography (EEG).
  Interventions: Behavioral: Behavioral Activation therapy; Behavioral: Computer-based behavioral assessment; Behavioral: Surveys and Interviews; Device: Magnetic resonance imaging (MRI); Device: Electroencephalography (EEG)

INTERVENTIONS:
Behavioral: Exposure-based therapy — Exposure-based therapy
  Arms: Exposure-based therapy
Behavioral: Behavioral Activation therapy — Behavioral Activation therapy
  Arms: Behavioral Activation therapy
Behavioral: Computer-based behavioral assessment — Computer-based tasks during which participants respond to images on the screen, including abstract images, emotional faces, and pleasant and unpleasant images.
Behavioral: Surveys and Interviews — Surveys and interviews in which participants will be asked to answer questions related to their mental and physical health history and current symptoms.
Device: Magnetic resonance imaging (MRI) — Magnetic resonance imaging (MRI) will be used to obtain information concerning the structure of the brain, as well as to assess changes associated with blood flow in the brain while participants are completing behavioral tasks (see description of computer-based behavioral assessment intervention).
Device: Electroencephalography (EEG) — Electroencephalography (EEG) will be used to assess changes in the electrical activity of the brain while participants are completing behavioral tasks (see description of computer-based behavioral assessment intervention).

SUMMARY:
This project aims to identify brain and behavioral characteristics of individuals experiencing symptoms of generalized anxiety disorder that will predict the effectiveness of Exposure-based therapy versus Behavioral Activation Therapy. Brain imaging aspects of the study will use functional magnetic resonance imaging (fMRI) and electroencephalography (EEG). Behavioral assessments will include self-report questionnaires, computer-based and observational tasks, and interviews. Assessments will focus on how individuals process positive information (such as reward) and negative information (such as distressing images), as well as how people make decisions. These assessments will be conducted across 2-3 in-person sessions prior to beginning the treatment, and will be repeated across 2-3 in-person sessions after completing treatment. A blood draw will also be conducted pre- and post- treatment. Both the Exposure-based and Behavior Activation therapy will consist of 10, 90-minute weekly therapy sessions conducted in small groups.

DETAILED DESCRIPTION:
Generalized anxiety disorder (GAD) is the most common anxiety disorder in primary care, with lifetime prevalence rates of 6%. GAD leads to significant individual and socioeconomic burden (e.g., due to days lost at work and increased health care utilization). Although there is significant comorbidity with major depressive disorder (MDD), a GAD diagnosis conveys a much poorer prognosis, with only 58% with GAD vs. 80% with MDD alone obtaining remission in two years. This highlights the importance of effectively treating GAD, for improving mental and physical health and decreasing socioeconomic burden. First-line treatments include medication (e.g., selective serotonin reuptake inhibitors [SSRIs]) and psychotherapy (e.g., cognitive behavioral therapy [CBT]). While both are superior to placebo, only 40-60% experience significant improvement, with at least 25% relapsing within a year. Thus, long-lasting improvements are occurring in less than 50% of patients. This ineffectiveness has been moderately associated with symptom severity, illness duration, and comorbidity, but these findings do not provide any strategies for improving treatment effectiveness. The current study will seek to identify behavioral or cognitive-affective predictors that indicate how well a patient is responding to treatment so that interventions can be further individualized to more effectively treat refractory patients.

The overall aim of this study are to identify whether neural, biological, and behavioral responses related to the arbitration of conflicting avoidance and approach drives can predict response to Exposure-based versus Behavioral Activate therapy for individuals with generalized anxiety disorder (with or without co-morbid major depressive disorder). This will be accomplished using behavioral, functional magnetic resonance imaging (fMRI), and genetic analyses pre and post Behavioral Activation therapy. Research subjects will include treatment-seeking individuals with clinically significant symptoms of unipolar depression. Diagnosis will be assessed using structured clinical interviews. Anxious and depressive symptom severity, personality characteristics, and general functioning will be collected via self-report paper-and-pencil questionnaires. Objective measures of approach, avoidance, and conflict behavioral responses will be collected using computer-administered testing and related neural responsivity will be measured using fMRI. For exploratory aims, a blood draw will be collect pre and post-treatment to examine genetic factors that may predict response to behavior therapy. This research has the potential to identify neural and behavioral approach-avoidance characteristics that can help predict which patients are likely to respond to Exposure-based versus Behavioral Activation therapy (i.e., predictors of treatment effectiveness) and reveal targets for future treatment modifications.

Aim 1: Examine relationships among approach-avoidance behavior and neural responses, and baseline GAD symptom severity.

Hypothesis 1.1: Approach and conflict arbitration behavior will explain significant variance in baseline symptoms above and beyond avoidance-related behavior.

Hypothesis 1.2: Approach (striatum) and conflict arbitration (lateral PFC) neural activity will explain significant variance in baseline symptoms above and beyond avoidance-related (amygdala) neural activity.

Aim 2: Examine how multi-level approach-avoidance behavior and neural responses predict individualized response to Exposure-based therapy for GAD (compared to Behavioral Activation).

Hypothesis 2.1: Approach-related and conflict arbitration behavior will help predict treatment response above and beyond avoidance-related behavior and baseline symptom severity.

Hypothesis 2.2: Activity in approach-related and conflict arbitration neural circuitry will predict treatment response above and beyond activity in avoidance-related neural circuitry.

Aim 3: Identify the changes in approach-avoidance processes that relate to Exposure therapy elicited functional improvement (compared to Behavioral Activation).

Hypothesis 3.1: The degree to which conflict arbitration abilities increase with treatment will positively relate to functional improvement from pre- to post-treatment.

The statistical analysis plan was described within a protocol paper published in 2020 (Santiago et al., 2020), which is cited in the References section.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18-55
2. All genders
3. All races
4. Eligibility as clinically significant anxiety will be determined by:

   * Scoring greater than 7 on the Overall Anxiety Severity and Impairment Scale (OASIS) or greater than 10 on the generalized anxiety disorder 7-item scale (GAD-7) and/or diagnosis of Generalized Anxiety Disorder.
   * Self-report that they are interested in obtaining treatment for anxiety.
   * Anxiety symptoms are the primary disorder of concern.
5. Able to provide written, informed consent
6. Have sufficient proficiency in English language to understand and complete interviews, questionnaires, and all other study procedures

Exclusion Criteria:

1. Has a history of unstable liver or renal insufficiency; glaucoma; significant and unstable cardiac, vascular, pulmonary, gastrointestinal, endocrine, neurologic, hematologic, rheumatologic, or metabolic disturbance; or any other condition that would make participation not be in the best interest (e.g., compromise the well-being) of the subject or that could prevent, limit, or confound the protocol-specified assessments.
2. A history of drug or alcohol abuse in the past 6 months,
3. Has any of the following diagnostic and statistical manual (DSM-5) disorders:

   * Schizophrenia Spectrum and Other Psychotic Disorders
   * Bipolar and Related Disorders
   * Obsessive-Compulsive and Related Disorders
   * Anorexia or Bulimia Nervosa
   * Substance use disorder within 6 months
4. Moderate to severe traumatic brain injury (>30 min. loss of consciousness or >24 hours posttraumatic amnesia) or other neurocognitive disorder with evidence of neurological deficits, neurological disorders, or severe or unstable medical conditions that might be compromised by participation in the study.
5. Active suicidal ideation with intent or plan
6. Current use of a medication that could affect brain functioning (e.g., anxiolytics, antipsychotics, mood stabilizers). However, participants reporting current use of prescribed antidepressants (selective serotonin reuptake inhibitors [SSRIs]) will be included as long as the dose has been stable for 6 weeks prior to enrolling in the study.
7. Prescription of a medication outside of the accepted range, as determined by the best clinical practices and current research
8. Taking drugs that affect the fMRI hemodynamic response.
9. MRI contraindications including: cardiac pacemaker, metal fragments in eyes/skin/body (shrapnel), aortic/aneurysm clips, prosthesis, by-pass surgery/coronary artery clips, hearing aid, heart valve replacement, shunt (ventricular or spinal), electrodes, metal plates/pins/screws/wires, or neuro/bio-stimulators (TENS unit), persons who have ever been a professional metal worker/welder, history of eye surgery/eyes washed out because of metal, vision problems uncorrectable with lenses, inability to lie still on one's back for 60-120 minutes; prior neurosurgery; tattoos or cosmetic makeup with metal dyes, unwillingness to remove body piercings, and pregnancy
10. Unwillingness or inability to complete any of the major aspects of the study protocol, including magnetic resonance imaging (i.e., due to claustrophobia), blood draws, or behavioral assessment. However, failing to complete some individual aspects of these assessment sessions will be acceptable (i.e., being unwilling to answer individual items on some questionnaires or being unwilling to complete a behavioral task)
11. Non-correctable vision or hearing problems
12. Report of severe depressive symptoms, as indicated by a score greater than 17 on the Patient Health Questionnaire 9-item (PHQ-9).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 121 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2021-07-27 (Actual); Study Completion 2022-03-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robin L Aupperle, Ph.D., Principal Investigator — Laureate Institute for Brain Research
Locations (1):
- Laureate Institute for Brain Research, Tulsa, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data may be made available to other individual researchers upon request to the principal investigator, Dr. Robin Aupperle.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Data may be available for sharing after a request is received. The duration of time in which that data is shared will be determined on a case by case basis.

REFERENCES:
- [Background] Cuijpers P, Sijbrandij M, Koole S, Huibers M, Berking M, Andersson G. Psychological treatment of generalized anxiety disorder: a meta-analysis. Clin Psychol Rev. 2014 Mar;34(2):130-40. doi: 10.1016/j.cpr.2014.01.002. Epub 2014 Jan 10. PMID 24487344
- [Background] Arch JJ, Ayers CR. Which treatment worked better for whom? Moderators of group cognitive behavioral therapy versus adapted mindfulness based stress reduction for anxiety disorders. Behav Res Ther. 2013 Aug;51(8):434-42. doi: 10.1016/j.brat.2013.04.004. Epub 2013 May 2. PMID 23747582
- [Background] Aupperle RL, Paulus MP. Neural systems underlying approach and avoidance in anxiety disorders. Dialogues Clin Neurosci. 2010;12(4):517-31. doi: 10.31887/DCNS.2010.12.4/raupperle. PMID 21319496
- [Background] Aupperle RL, Melrose AJ, Francisco A, Paulus MP, Stein MB. Neural substrates of approach-avoidance conflict decision-making. Hum Brain Mapp. 2015 Feb;36(2):449-62. doi: 10.1002/hbm.22639. Epub 2014 Sep 15. PMID 25224633
- [Background] Aupperle RL, Sullivan S, Melrose AJ, Paulus MP, Stein MB. A reverse translational approach to quantify approach-avoidance conflict in humans. Behav Brain Res. 2011 Dec 1;225(2):455-63. doi: 10.1016/j.bbr.2011.08.003. Epub 2011 Aug 6. PMID 21843556
- [Background] Santiago J, Akeman E, Kirlic N, Clausen AN, Cosgrove KT, McDermott TJ, Mathis B, Paulus M, Craske MG, Abelson J, Martell C, Wolitzky-Taylor K, Bodurka J, Thompson WK, Aupperle RL. Protocol for a randomized controlled trial examining multilevel prediction of response to behavioral activation and exposure-based therapy for generalized anxiety disorder. Trials. 2020 Jan 6;21(1):17. doi: 10.1186/s13063-019-3802-9. PMID 31907032
- [Derived] Berg H, McDermott TJ, Kuplicki R, Yeh HW, Thompson WK, Smith R, Akeman E, Kirlic N, Clausen A, Cannon M, White E, Martell CR, Wolitzky-Taylor KB, Craske MG, Abelson JL, Paulus MP, Aupperle RL. Prediction of generalized anxiety disorder treatment outcomes with neurobehavioral responses to approach-avoidance conflict: a randomized clinical trial. Transl Psychiatry. 2025 Jul 5;15(1):231. doi: 10.1038/s41398-025-03460-x. PMID 40617801
- [Derived] Berg H, Eun YJ, Yu X, McDermott TJ, Akeman E, Kuplicki R, Yeh HW, Thompson W, Martell CR, Wolitzky-Taylor KB, Craske MG, Paulus MP, Aupperle RL. Neural activity to reward and loss predicting treatment outcomes for adults with generalized anxiety disorder: A randomized clinical trial. J Mood Anxiety Disord. 2025 Mar;9:100107. doi: 10.1016/j.xjmad.2025.100107. Epub 2025 Jan 8. PMID 40384942
- [Derived] Berg H, Akeman E, McDermott TJ, Cosgrove KT, Kirlic N, Clausen A, Cannon M, Yeh HW, White E, Thompson WK, Choquette EM, Sturycz-Taylor CA, Cochran G, Ramirez S, Martell CR, Wolitzky-Taylor KB, Craske MG, Abelson JL, Paulus MP, Aupperle RL. A randomized clinical trial of behavioral activation and exposure-based therapy for adults with generalized anxiety disorder. J Mood Anxiety Disord. 2023 Jun;1:100004. doi: 10.1016/j.xjmad.2023.100004. Epub 2023 Jun 9. PMID 38384390

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: After enrollment, participants completed baseline assessments prior to being randomized to a treatment arm. A total of 121 were rolled in the study. Prior to randomization, 27 participants withdrew from the study due to no longer meeting criteria (N=9), indicated being no longer interested in participating (N=8), and other or unknown reasons (N=10), leaving N=94 being randomized and starting treatment.
Groups:
- Exposure-based Therapy: Participants will complete 10, 90-minute sessions of Exposure-based therapy, conducted using a group format. Each group will include 8-12 participants. Exposure-based therapy seeks to increase abilities to manage anxiety through repeated practice in facing the situations or thoughts that are the focus of worry or fear.
- Behavioral Activation Therapy: Participants will complete 10, 90-minute sessions of Behavioral Activation therapy, conducted using a group format. Each group will include 8-12 participants. Behavioral Activation therapy seeks to target behaviors that might maintain or worsen negative mood.
Period: Overall Study
Arm/Group | Exposure-based Therapy | Behavioral Activation Therapy
Started | 46 | 48
Completed | 32 (Completion defined as attending at least 7 sessions of therapy.) | 38 (Completion defined as attending at least 7 sessions of therapy.)
Not Completed | 14 | 10
Not completed — Withdrawal by Subject | 14 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Exposure-based Therapy | Behavioral Activation Therapy | Total
Number analyzed (Participants) | 46 | 48 | 94
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 46 | 48 | 94
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.96 (10.63) | 34.27 (10.54) | 34.61 (10.53)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44 | 38 | 82
  Male | 2 | 10 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 4
  Not Hispanic or Latino | 44 | 46 | 90
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 9 | 11 | 20
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 6 | 7
  White | 30 | 27 | 57
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 4 | 3 | 7
Region of Enrollment [Number; unit: participants]
  United States | 46 | 48 | 94
Education [Count of Participants; unit: Participants]
  Less than high school | 1 | 1 | 2
  High school or GED | 4 | 4 | 8
  Some college, no degree | 12 | 14 | 26
  Bachelor's degree | 10 | 16 | 26
  Associate's degree | 4 | 3 | 7
  Master's degree | 13 | 10 | 23
  Professional / doctoral degree | 2 | 0 | 2
GAD7 Baseline Score [Mean (Standard Deviation); unit: units on a scale] — Baseline Generalized Anxiety Disorder Symptoms as Measured by the self-report measure, the Generalized Anxiety Disorder - 7 Item Scale (GAD-7). Scores on the Generalized Anxiety Disorder - 7 item scale (GAD-7) range from 0 to 21, higher scores reflect greater symptom severity.
  units on a scale | 12.93 (4.62) | 11.30 (3.73) | 12.12 (4.25)

OUTCOME MEASURES:

1. Primary Outcome: For Aim1: Baseline Generalized Anxiety Disorder Symptoms as Measured by the Generalized Anxiety Disorder - 7 Item Scale (GAD-7).
Description: Test the relationship between imaging and behavioral factors and the level of symptoms at baseline assessment. Scores on the Generalized Anxiety Disorder - 7 item scale (GAD-7) range from 0 to 21, higher scores reflect greater symptom severity.
Time Frame: Baseline assessment (one time point)
Population: Participants who 1) had usable pre-treatment fMRI data and 2) completed treatment with at least 7 sessions attended
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Exposure-based Therapy | Behavioral Activation Therapy
Number analyzed (Participants) | 27 | 30
units on a scale | 12.85 (5.33) | 11.62 (3.38)
Statistical Analysis 1: Comparison: Exposure-based Therapy vs Behavioral Activation Therapy; Test type: Other — Correlation between conflict approach behavior and GAD-7 scores at baseline; p = .088, Pearson correlation; Pearson correlation = 0.23
Statistical Analysis 2: Comparison: Exposure-based Therapy vs Behavioral Activation Therapy; Correlation of baseline response time during conflict with baseline GAD-7 scores; Test type: Other; p = .134, Pearson correlation; Pearson correlation = -0.2
Statistical Analysis 3: Comparison: Exposure-based Therapy vs Behavioral Activation Therapy; Correlation of baseline striatum response to points (reward) with baseline GAD-7 scores; Test type: Other; p = .032, Pearson correlation; Pearson correlation = .12
Statistical Analysis 4: Comparison: Exposure-based Therapy vs Behavioral Activation Therapy; Correlation of baseline right amygdala activity during negative images with baseline GAD7 scores; Test type: Other; p = 0.375, Pearson correlation; Pearson correlation = -0.12
Statistical Analysis 5: Comparison: Exposure-based Therapy vs Behavioral Activation Therapy; Correlation of baseline right dlPFC activity during conflict decision-making with baseline GAD-7 scores; Test type: Other; p = .651, Pearson correlation; Pearson correlation = 0.06
Statistical Analysis 6: Comparison: Exposure-based Therapy vs Behavioral Activation Therapy; Test type: Other — Correlation of baseline striatum response to negative pictures with baseline GAD-7 scores; p = .008, Pearson correlation; Pearson correlation = -0.35

2. Primary Outcome: For Aims 2 and 3: Change in Generalized Anxiety Disorder Symptoms as Measured by the Generalized Anxiety Disorder - 7 Item Scale (GAD-7).
Description: Test the predictive effects of imaging and behavioral factors on change in symptoms at baseline compared to within 6 weeks after completing treatment. Scores on the Generalized Anxiety Disorder - 7 item scale (GAD-7) range from 0 to 21, higher scores reflect greater symptom severity.
Time Frame: Trajectory of change from pre- to post- treatment; last time point assessed within 6 weeks following last treatment session, on average at 16 weeks after baseline assessment.
Population: Participants who had usable baseline fMRI data and completed treatment. Outcome measure data entered for post-treatment timepoint or last timepoint collected.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Exposure-based Therapy | Behavioral Activation Therapy
Number analyzed (Participants) | 27 | 29
units on a scale | 8.48 (4.20) | 5.90 (3.97)
Statistical Analysis 1: Comparison: Exposure-based Therapy vs Behavioral Activation Therapy; Assess left amygdala response to positive picture decision outcomes as a predictor of GAD-7 symptom improvement: time x L. Amyg x treatment-arm interaction; Test type: Other; p = .007, Regression, Linear — The a priori threshold for statistical significance after Bonferroni correction for multiple comparisons was p<.0071; Slope = -1.51, 95% CI 2-sided [-2.62 to -0.41] — Those with lower levels of baseline left amygdala response to positive picture outcomes had favorable GAD symptom improvements in BA and limited GAD symptom improvements in EXP
Statistical Analysis 2: Comparison: Exposure-based Therapy vs Behavioral Activation Therapy; Baseline approach behavior during conflict trials predicting trajectory of GAD-7 symptoms: time main effect; Test type: Other; p = 0.238, Regression, Linear; Slope = 0.36, 95% CI 2-sided [-0.24 to 0.97]
Statistical Analysis 3: Comparison: Exposure-based Therapy vs Behavioral Activation Therapy; Relationship between baseline approach behavior on conflict trials and the trajectory of GAD-7 symptoms: time x treatment interaction effect; Test type: Superiority; p = .262, Regression, Linear; Slope = -0.49, 95% CI 2-sided [-1.36 to 0.37]
Statistical Analysis 4: Comparison: Exposure-based Therapy vs Behavioral Activation Therapy; relationship between baseline response time on conflict trials and trajectory of GAD-7 symptoms: time main effects; Test type: Other; p = .222, Regression, Linear; Slope = 2.37, 95% CI 2-sided [-1.44 to 6.19]
Statistical Analysis 5: Comparison: Exposure-based Therapy vs Behavioral Activation Therapy; Relationship between baseline average RT during conflict trials on the AAC and trajectory of GAD-7 symptoms: time x treatment interaction effect; Test type: Superiority; p = .942, Regression, Linear; Slope = -0.23, 95% CI 2-sided [-6.48 to 6.02]
Statistical Analysis 6: Comparison: Exposure-based Therapy vs Behavioral Activation Therapy; Relationship of striatum activity during points outcomes (reward) with GAD-7 trajectory: time main effects; Test type: Other; p = .932, Regression, Linear; Slope = -0.05, 95% CI 2-sided [-1.2 to 1.1]
Statistical Analysis 7: Comparison: Exposure-based Therapy vs Behavioral Activation Therapy; Relationship of striatum activity during points outcomes (reward) with GAD-7 trajectory: time x treatment interaction effects; Test type: Superiority; p = .922, Regression, Linear; Slope = -0.08, 95% CI 2-sided [-1.7 to 1.53]
Statistical Analysis 8: Comparison: Exposure-based Therapy vs Behavioral Activation Therapy; Relationship of right amygdala activity during negative images with GAD-7 trajectory: time main effects; Test type: Other; p = .998, Regression, Linear; Slope = 0.00, 95% CI 2-sided [-.99 to .99]
Statistical Analysis 9: Comparison: Exposure-based Therapy vs Behavioral Activation Therapy; Relationship of right amygdala activity during negative images with GAD-7 trajectory: time x treatment interaction; Test type: Superiority; p = .234, Regression, Linear; Slope = -0.88, 95% CI 2-sided [-2.34 to .57]
Statistical Analysis 10: Comparison: Exposure-based Therapy vs Behavioral Activation Therapy; Relationship of right dlPFC activity during conflict decisions with GAD-7 trajectory: time main effects; Test type: Other; p = .967, Regression, Linear; Slope = -0.03, 95% CI 2-sided [-1.53 to 1.47]
Statistical Analysis 11: Comparison: Exposure-based Therapy vs Behavioral Activation Therapy; Relationship of right dlPFC activity during conflict decision-making with GAD-7 trajectory: time x treatment interaction effect; Test type: Other; p = 0.504, Regression, Linear; Slope = 0.74, 95% CI 2-sided [-1.43 to 2.91]
Statistical Analysis 12: Comparison: Exposure-based Therapy vs Behavioral Activation Therapy; Change in conflict arbitration (AAC conflict RTpost-RTpre) predicting trajectories of GAD-7 scores over the 10 sessions: Time x RT_Change interaction; Test type: Other; p = 0.612, Regression, Linear; Slope = -1.68, 95% CI 2-sided [-8.21 to 4.84]
Statistical Analysis 13: Comparison: Exposure-based Therapy vs Behavioral Activation Therapy; change in conflict arbitration response time (AAC conflict RTpost-RTpre) predicting trajectories of GAD-7 scores over 10 sessions: RT_Change x Time x Treatment interaction; Test type: Superiority; p = .259, Regression, Linear; Slope = 5.08, 95% CI 2-sided [-3.76 to 13.92]
Statistical Analysis 14: Comparison: Exposure-based Therapy vs Behavioral Activation Therapy; Change in behavior (AAC conflict post-pre) in predicting trajectories of GAD-7 scores over the 10 sessions: Time x Behavior_change interaction; Test type: Other; p = .209, Regression, Linear; Slope = -0.53, 95% CI 2-sided [-1.35 to 0.30]
Statistical Analysis 15: Comparison: Exposure-based Therapy vs Behavioral Activation Therapy; Change in behavior (AAC conflict post-pre) in predicting trajectories of GAD-7 scores over the 10 sessions: Time x Behavior_change x Treatment interaction; Test type: Superiority; p = 0.013, Regression, Linear; Slope = 1.53, 95% CI 2-sided [0.33 to 2.73]

3. Secondary Outcome: Change in Anxiety Symptoms as Measured by the Patient Reported Outcomes Measurement Information System (PROMIS) Anxiety Scale.
Description: Test the predictive effects of imaging and behavioral factors on change in symptoms at baseline compared to within 6 weeks after completing treatment. The PROMIS Anxiety Scale yields t-scores, higher scores indicate greater symptom severity, with 50 indicating the population mean and a standard deviation of 10.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Exposure-based Therapy | Behavioral Activation Therapy
Number analyzed (Participants) | 27 | 29
T-score | 60.68 (5.86) | 55.98 (7.23)
Statistical Analysis 1: Comparison: Exposure-based Therapy vs Behavioral Activation Therapy; Baseline emotional conflict, a computational parameter reflecting avoidance relative to reward value, as a predictor of the linear trajectory of symptom change over time: time x EC interaction; Test type: Other; p = 0.006, Regression, Linear — The a priori threshold for statistical significance after Bonferroni correction for multiple comparisons was p<.0125; Slope = -2.95, 95% CI 2-sided [-5.06 to -0.84]
Statistical Analysis 2: Comparison: Exposure-based Therapy vs Behavioral Activation Therapy; Assess avoidance behavior on conflict trials as a predictor of PROMIS Anxiety symptom improvement: time x avoidance interaction; Test type: Other; p = 0.003, Regression, Linear; Slope = -1.02, 95% CI 2-sided [-1.68 to -0.36]
Statistical Analysis 3: Comparison: Exposure-based Therapy vs Behavioral Activation Therapy; Assess left dlPFC response to baseline negative picture decision outcomes as a predictor of PROMIS Anxiety symptom improvement: time x L. dlPFC interaction; Test type: Other; p = .007, Regression, Linear — The a priori threshold for statistical significance after Bonferroni correction for multiple comparisons was p<.0071; Slope = -1.88, 95% CI 2-sided [-2.89 to -0.87]
Statistical Analysis 4: Comparison: Exposure-based Therapy vs Behavioral Activation Therapy; Relationships between baseline average approach behavior during conflict trials on the AAC and trajectory of PROMIS Anxiety symptoms; Test type: Other; p = .003, Regression, Linear; Slope = 1.02, 95% CI 2-sided [0.36 to 1.68]
Statistical Analysis 5: Comparison: Exposure-based Therapy vs Behavioral Activation Therapy; Relationships between baseline average approach behavior during conflict trials on the AAC and trajectory of PROMIS Anxiety symptoms: time x treatment x approach behavior interaction; Test type: Superiority; p = .258, Regression, Linear; Slope = -0.54, 95% CI 2-sided [-1.48 to 0.4]
Statistical Analysis 6: Comparison: Exposure-based Therapy vs Behavioral Activation Therapy; Relationships between baseline average RT during conflict trials on the AAC and trajectory of PROMIS Anxiety symptoms: time x approach behavior interaction; Test type: Other; p = .56, Regression, Linear; Slope = 1.3, 95% CI 2-sided [-3.08 to 5.69]
Statistical Analysis 7: Comparison: Exposure-based Therapy vs Behavioral Activation Therapy; Relationships between baseline average RT (response time) during conflict trials on the AAC and trajectory of PROMIS Anxiety symptoms: time x treatment x RT interaction; Test type: Superiority; p = .629, Regression, Linear; Slope = -1.77, 95% CI 2-sided [-8.95 to 5.41]
Statistical Analysis 8: Comparison: Exposure-based Therapy vs Behavioral Activation Therapy; Relationship of striatum activity during points outcomes (reward) with PROMIS ANXIETY trajectory: time x striatum interaction effects; Test type: Other; p = 0.75, Regression, Linear; Slope = -0.21, 95% CI 2-sided [-1.51 to 1.09]
Statistical Analysis 9: Comparison: Exposure-based Therapy vs Behavioral Activation Therapy; Relationship of striatum activity during points outcomes (reward) with PROMIS Anxiety trajectory: time x treatment x striatum interaction effects; Test type: Superiority; p = .169, Regression, Linear; Slope = 1.27, 95% CI 2-sided [-0.54 to 3.09]
Statistical Analysis 10: Comparison: Exposure-based Therapy vs Behavioral Activation Therapy; Relationship of right amygdala activity during negative images with PROMIS Anxiety trajectory: time x amygdala interaction; Test type: Other; p = 0.792, Regression, Linear; Slope = 0.15, 95% CI 2-sided [-1.00 to 1.31]
Statistical Analysis 11: Comparison: Exposure-based Therapy vs Behavioral Activation Therapy; Relationship of right amygdala activity during negative images with PROMIS Anxiety trajectory: time x treatment amygdala interaction; Test type: Superiority; p = .396, Regression, Linear; Slope = -0.73, 95% CI 2-sided [-2.41 to 0.96]
Statistical Analysis 12: Comparison: Exposure-based Therapy vs Behavioral Activation Therapy; Relationship of right dlPFC activity during negative images with PROMIS Anxiety trajectory: time x dlPFC interaction; Test type: Other; p = .009, Regression, Linear; Slope = -1.55, 95% CI 2-sided [-2.7 to -0.4]
Statistical Analysis 13: Comparison: Exposure-based Therapy vs Behavioral Activation Therapy; Relationship of right dlPFC activity during negative images with PROMIS Anxiety trajectory: time x treatment dlPFC interaction; Test type: Superiority; p = 0.724, Regression, Linear; Slope = 0.28, 95% CI 2-sided [-1.28 to 1.84]
Statistical Analysis 14: Comparison: Exposure-based Therapy vs Behavioral Activation Therapy; Change in conflict arbitration response time (AAC conflict RT post-pre) predicting trajectories of GAD-7 scores over the 10 sessions: Time x RT_change interaction; Test type: Other; p = .209, Regression, Linear; Slope = -4.99, 95% CI 2-sided [-12.79 to 2.80]
Statistical Analysis 15: Comparison: Exposure-based Therapy vs Behavioral Activation Therapy; Change in conflict arbitration response time (AAC conflict RT post-pre) predicting trajectories of GAD-7 scores over the 10 sessions: Time x Treatment x RT_change interaction; Test type: Superiority; p = 0.017, Regression, Linear; Slope = 12.68, 95% CI 2-sided [2.23 to 23.13]
Statistical Analysis 16: Comparison: Exposure-based Therapy vs Behavioral Activation Therapy; Change in behavior (AAC conflict post-pre) predicting trajectories of GAD-7 scores over the 10 sessions: Time x Behavior_change interaction; Test type: Other; p = .259, Regression, Linear; Slope = -0.58, 95% CI 2-sided [-1.59 to 0.43]
Statistical Analysis 17: Comparison: Exposure-based Therapy vs Behavioral Activation Therapy; Change in behavior (AAC conflict post-pre) predicting trajectories of GAD-7 scores over the 10 sessions: Time x Treatment x Behavior_change interaction; Test type: Other; p = .150, Regression, Linear; Slope = 1.07, 95% CI 2-sided [-0.39 to 2.54]

4. Secondary Outcome: Change in Depressive Symptoms as Measured by the Patient Reported Outcomes Measurement Information System (PROMIS) Depression Scale.
Description: Test the predictive effects of imaging and behavioral factors on change in symptoms at baseline compared to within 6 weeks after completing treatment. The PROMIS Depression scale yields t-scores; higher scores indicate greater symptom severity, with population mean being 50 and standard deviation of 10.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Exposure-based Therapy | Behavioral Activation Therapy
Number analyzed (Participants) | 27 | 29
T-score | 53.70 (6.87) | 52.12 (4.73)
Statistical Analysis 1: Comparison: Exposure-based Therapy vs Behavioral Activation Therapy; Assess emotional conflict, a computational parameter reflecting avoidance relative to reward value, as a predictor of PROMIS Depression scores. Time x EC interaction; Test type: Other; p = 0.001, Regression, Linear — The a priori threshold for statistical significance after Bonferroni correction for multiple comparisons was p<.0125; Slope = -3.52, 95% CI 2-sided [-5.57 to -1.47]
Statistical Analysis 2: Comparison: Exposure-based Therapy vs Behavioral Activation Therapy; Baseline left dlPFC response to negative pictures as a predictor of PROMIS depression symptom improvement: time x L. dlFPC interaction; Test type: Other; p < .001, Regression, Linear — The a priori threshold for statistical significance after Bonferroni correction for multiple comparisons was p<.0125; Slope = -1.93, 95% CI 2-sided [-2.91 to -0.95]
Statistical Analysis 3: Comparison: Exposure-based Therapy vs Behavioral Activation Therapy; Baseline striatum response to monetary outcomes as a predictor of improvement in depressive symptoms: time x treatment x striatum interaction; Test type: Other; p = .036, Regression, Linear — Threshold for statistical significance is 0.05; Slope = -2.02, 95% CI 2-sided [-3.9 to -0.13]
Statistical Analysis 4: Comparison: Exposure-based Therapy vs Behavioral Activation Therapy; Relationships between baseline average approach behavior during conflict trials on the AAC and trajectory of PROMIS Depression symptoms: time x approach behavior interaction; Test type: Other; p < .001, Regression, Linear — The a priori threshold for statistical significance after Bonferroni correction for multiple comparisons was p<.0125; Slope = -1.21, 95% CI 2-sided [-1.85 to -0.58]
Statistical Analysis 5: Comparison: Exposure-based Therapy vs Behavioral Activation Therapy; Relationships between baseline average approach behavior during conflict trials on the AAC and trajectory of PROMIS Depression symptoms: time x treatment x approach behavior interaction; Test type: Superiority; p = .049, Regression, Linear; Slope = -0.91, 95% CI 2-sided [-1.81 to 0.00]
Statistical Analysis 6: Comparison: Exposure-based Therapy vs Behavioral Activation Therapy; Relationships between baseline average RT during conflict trials on the AAC and trajectory of PROMIS Depression symptoms: time x RT interaction; Test type: Other; p = .778, Regression, Linear; Slope = .6, 95% CI 2-sided [-3.6 to 4.81]
Statistical Analysis 7: Comparison: Exposure-based Therapy vs Behavioral Activation Therapy; Relationships between baseline average RT during conflict trials on the AAC and trajectory of PROMIS Depression symptoms: time x treatment x RT interaction; Test type: Superiority; p = .696, Regression, Linear; Slope = 1.38, 95% CI 2-sided [-5.56 to 8.31]
Statistical Analysis 8: Comparison: Exposure-based Therapy vs Behavioral Activation Therapy; Relationship of striatum activity during points outcomes (reward) with PROMIS Depression trajectory: time x striatum interaction effects; Test type: Other; p = .503, Regression, Linear; Slope = .44, 95% CI 2-sided [-0.84 to 1.71]
Statistical Analysis 9: Comparison: Exposure-based Therapy vs Behavioral Activation Therapy; Relationship of right amygdala activity during negative images with PROMIS Depression trajectory: time x amygdala interaction; Test type: Other; p = .114, Regression, Linear; Slope = -0.9, 95% CI 2-sided [-2.02 to .22]
Statistical Analysis 10: Comparison: Exposure-based Therapy vs Behavioral Activation Therapy; Relationship of right amygdala activity during negative images with PROMIS Depression trajectory: time x treatment amygdala interaction; Test type: Superiority; p = .561, Regression, Linear; Slope = 0.48, 95% CI 2-sided [-1.15 to 2.11]
Statistical Analysis 11: Comparison: Exposure-based Therapy vs Behavioral Activation Therapy; Relationship of right dlPFC activity during negative images with PROMIS Depression trajectory: time x dlPFC interaction; Test type: Other; p = .007, Regression, Linear; Slope = -1.54, 95% CI 2-sided [-2.66 to -0.42]
Statistical Analysis 12: Comparison: Exposure-based Therapy vs Behavioral Activation Therapy; Relationship of right dlPFC activity during negative images with PROMIS Depression trajectory: time x treatment dlPFC interaction; Test type: Superiority; p = 0.403, Regression, Linear; Slope = 0.65, 95% CI 2-sided [-0.87 to 2.17]
Statistical Analysis 13: Comparison: Exposure-based Therapy vs Behavioral Activation Therapy; [analysis description as in outcome 3, analysis 14]; Test type: Other; p = 0.681, Regression, Linear; Slope = -1.51, 95% CI 2-sided [-8.76 to 5.73]
Statistical Analysis 14: Comparison: Exposure-based Therapy vs Behavioral Activation Therapy; [analysis description as in outcome 3, analysis 15]; Test type: Superiority; p = .264, Regression, Linear; Slope = 5.61, 95% CI 2-sided [-4.24 to 15.46]
Statistical Analysis 15: Comparison: Exposure-based Therapy vs Behavioral Activation Therapy; [analysis description as in outcome 3, analysis 16]; Test type: Other; p = .367, Regression, Linear; Slope = -0.43, 95% CI 2-sided [-1.38 to 0.51]
Statistical Analysis 16: Comparison: Exposure-based Therapy vs Behavioral Activation Therapy; [analysis description as in outcome 3, analysis 17]; Test type: Other; p = .211, Regression, Linear; Slope = 0.88, 95% CI 2-sided [-0.50 to 2.25]

5. Secondary Outcome: Change in Level of Disability as Measured by the Sheehan Disability Scale
Description: Test the predictive effects of imaging and behavioral factors on change in symptoms at baseline compared to within 6 weeks after completing treatment. The Sheehan Disability Scale assesses functional impairment in the domains of work/school, social life, and family life. Participants are provided with a 0-10 visual analog scale with spatiovisual, numeric, and descriptive anchors and asked to rate the extent to which their symptoms have interfered with their functioning on each item for total score ranges of 0-30. Higher scores indicate greater impairment.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Exposure-based Therapy | Behavioral Activation Therapy
Number analyzed (Participants) | 27 | 29
score on a scale | 8.93 (6.11) | 5.36 (5.47)
Statistical Analysis 1: Comparison: Exposure-based Therapy vs Behavioral Activation Therapy; Relationships between baseline average approach behavior during conflict trials on the AAC and trajectory of SDS score: time x approach behavior interaction; Test type: Other; p = 0.028, Regression, Linear; Slope = 0.74, 95% CI 2-sided [0.08 to 1.41]
Statistical Analysis 2: Comparison: Exposure-based Therapy vs Behavioral Activation Therapy; Relationships between baseline average approach behavior during conflict trials on the AAC and trajectory of SDS symptoms: time x treatment x approach behavior interaction; Test type: Superiority; p = 0.251, Regression, Linear; Slope = -0.55, 95% CI 2-sided [-1.49 to 0.39]
Statistical Analysis 3: Comparison: Exposure-based Therapy vs Behavioral Activation Therapy; Relationships between baseline average RT during conflict trials on the AAC and trajectory of SDS symptoms: time x RT interaction; Test type: Other; p = 0.902, Regression, Linear; Slope = -0.26, 95% CI 2-sided [-4.49 to 3.96]
Statistical Analysis 4: Comparison: Exposure-based Therapy vs Behavioral Activation Therapy; Relationships between baseline average RT during conflict trials on the AAC and trajectory of SDS symptoms: time x treatment x RT interaction; Test type: Superiority; p = .519, Regression, Linear; Slope = 2.23, 95% CI 2-sided [-4.55 to 9.01]
Statistical Analysis 5: Comparison: Exposure-based Therapy vs Behavioral Activation Therapy; Relationship of striatum activity during points outcomes (reward) with SDS trajectory: time x striatum interaction effects; Test type: Other; p = .326, Regression, Linear; Slope = -0.64, 95% CI 2-sided [-1.92 to 0.64]
Statistical Analysis 6: Comparison: Exposure-based Therapy vs Behavioral Activation Therapy; Relationship of striatum activity during points outcomes (reward) with SDS trajectory: time x treatment x striatum interaction effects; Test type: Superiority; p = .168, Regression, Linear; Slope = 1.26, 95% CI 2-sided [-0.53 to 3.05]
Statistical Analysis 7: Comparison: Exposure-based Therapy vs Behavioral Activation Therapy; Relationship of right amygdala activity during negative images with SDS trajectory: time x amygdala interaction; Test type: Other; p = .248, Regression, Linear; Slope = -0.50, 95% CI 2-sided [-1.34 to 0.35]
Statistical Analysis 8: Comparison: Exposure-based Therapy vs Behavioral Activation Therapy; Relationship of right amygdala activity during negative images with SDS trajectory: time x treatment amygdala interaction; Test type: Superiority; p = 0.603, Regression, Linear; Slope = 0.30, 95% CI 2-sided [-0.84 to 1.44]
Statistical Analysis 9: Comparison: Exposure-based Therapy vs Behavioral Activation Therapy; Relationship of right dlPFC activity during negative images with SDS trajectory: time x dlPFC interaction; Test type: Other; p = .107, Regression, Linear; Slope = -0.85, 95% CI 2-sided [-1.89 to 0.18]
Statistical Analysis 10: Comparison: Exposure-based Therapy vs Behavioral Activation Therapy; Relationship of right dlPFC activity during negative images with SDS trajectory: time x treatment x dlPFC interaction; Test type: Superiority; p = 0.846, Regression, Linear; Slope = 0.16, 95% CI 2-sided [-1.47 to 1.80]
Statistical Analysis 11: Comparison: Exposure-based Therapy vs Behavioral Activation Therapy; Change in conflict arbitration response time (AAC conflict RT post-pre) predicting trajectories of SDS scores over the 10 sessions: Time x RT_change interaction; Test type: Other; p = .561, Regression, Linear; Slope = -2.26, 95% CI 2-sided [-9.89 to 5.37]
Statistical Analysis 12: Comparison: Exposure-based Therapy vs Behavioral Activation Therapy; Change in conflict arbitration response time (AAC conflict RT post-pre) predicting trajectories of SDS scores over the 10 sessions: Time x Treatment x RT_change interaction; Test type: Superiority; p = .297, Regression, Linear; Slope = 5.45, 95% CI 2-sided [-4.80 to 15.70]
Statistical Analysis 13: Comparison: Exposure-based Therapy vs Behavioral Activation Therapy; Change in behavior (AAC conflict post-pre) predicting trajectories of SDS cores over the 10 sessions: Time x Behavior_change interaction; Test type: Other; p = .712, Regression, Linear; Slope = -0.18, 95% CI 2-sided [-1.15 to 0.79]
Statistical Analysis 14: Comparison: Exposure-based Therapy vs Behavioral Activation Therapy; Change in behavior (AAC conflict post-pre) predicting trajectories of SDS scores over the 10 sessions: Time x Treatment x Behavior_change interaction; Test type: Superiority; p = 0.431, Regression, Linear; Slope = 0.56, 95% CI 2-sided [-0.84 to 1.97]

6. Secondary Outcome: Worry Symptoms as Measured by the Penn State Worry Questionnaire
Description: Test the predictive effects of imaging and behavioral factors on post-treatment symptoms (within 6 weeks after completing treatment), covarying for baseline symptom severity. The PSWQ is a 16-item self-report scale designed to measure the trait of worry in adults. Scores range from 16 to 80 with higher scores indicative of higher levels of trait worry. Scores of 66 or greater are thought to indicate clinically significant worry.
Time Frame: Post- treatment; last time point assessed within 6 weeks following last treatment session, on average at 16 weeks after baseline assessment
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Exposure-based Therapy | Behavioral Activation Therapy
Number analyzed (Participants) | 27 | 29
score on a scale | 64.26 (10.29) | 56.29 (10.59)
Statistical Analysis 1: Comparison: Exposure-based Therapy vs Behavioral Activation Therapy; Relationships between baseline average approach behavior during conflict trials on the AAC and post-treatment PSWQ score: approach behavior main effect; Test type: Other; p = .276, Regression, Linear; Slope = -6.42, 95% CI 2-sided [-18.15 to 5.30]
Statistical Analysis 2: Comparison: Exposure-based Therapy vs Behavioral Activation Therapy; Relationships between baseline average approach behavior during conflict trials on the AAC and post-treatment PSWQ score: treatment x approach behavior interaction; Test type: Superiority; p = .520, Regression, Linear; Slope = 5.69, 95% CI 2-sided [-12.12 to 23.50]
Statistical Analysis 3: Comparison: Exposure-based Therapy vs Behavioral Activation Therapy; Relationships between baseline average RT during conflict trials on the AAC and trajectory of PSWQ score: RT main effect; Test type: Other; p = .199, Regression, Linear; Slope = -50.00, 95% CI 2-sided [-127.65 to 27.65]
Statistical Analysis 4: Comparison: Exposure-based Therapy vs Behavioral Activation Therapy; Relationships between baseline average RT during conflict trials on the AAC and trajectory of PSWQ score: treatment x RT interaction; Test type: Superiority; p = .191, Regression, Linear; Slope = 93.87, 95% CI 2-sided [-4.14 to 236.88]
Statistical Analysis 5: Comparison: Exposure-based Therapy vs Behavioral Activation Therapy; Relationship of striatum activity during points outcomes (reward) with PSWQ trajectory: striatum main effect; Test type: Other; p = 0.021, Regression, Linear; Slope = 27.35, 95% CI 2-sided [4.45 to 50.26]
Statistical Analysis 6: Comparison: Exposure-based Therapy vs Behavioral Activation Therapy; Relationship of striatum activity during points outcomes (reward) with PSWQ post-treatment: treatment x striatum interaction effects; Test type: Superiority; p = .734, Regression, Linear; Slope = -5.47, 95% CI 2-sided [-37.94 to 27.00]
Statistical Analysis 7: Comparison: Exposure-based Therapy vs Behavioral Activation Therapy; Relationship of right amygdala activity during negative images with PSWQ post-treatment: amygdala main effect; Test type: Other; p = .231, Regression, Linear; Slope = -9.79, 95% CI 2-sided [-26.11 to 6.53]
Statistical Analysis 8: Comparison: Exposure-based Therapy vs Behavioral Activation Therapy; Relationship of right amygdala activity during negative images with PSWQ post-treatment: treatment amygdala interaction; Test type: Superiority; p = .602, Regression, Linear; Slope = 8.55, 95% CI 2-sided [-24.48 to 41.58]
Statistical Analysis 9: Comparison: Exposure-based Therapy vs Behavioral Activation Therapy; Relationship of right dlPFC activity during negative images with PSWQ post-treatment: dlPFC main effect; Test type: Other; p = .369, Regression, Linear; Slope = -19.29, 95% CI 2-sided [-62.07 to 23.68]
Statistical Analysis 10: Comparison: Exposure-based Therapy vs Behavioral Activation Therapy; Relationship of right dlPFC activity during negative images with PSWQ post-treatment: treatment x dlPFC interaction; Test type: Superiority; p = .684, Regression, Linear; Slope = 9.12, 95% CI 2-sided [-36.05 to 54.29]
Statistical Analysis 11: Comparison: Exposure-based Therapy vs Behavioral Activation Therapy; Change in behavior (AAC conflict post-pre) predicting trajectories of PSWQ cores over the 10 sessions: Behavior_change main effect; Test type: Other; p = .487, Regression, Linear; Slope = 9.6, 95% CI 2-sided [-18.39 to 37.59]
Statistical Analysis 12: Comparison: Exposure-based Therapy vs Behavioral Activation Therapy; Change in behavior (AAC conflict post-pre) predicting trajectories of PSWQ scores over the 10 sessions: Treatment x Behavior_change interaction; Test type: Superiority; p = .033, Regression, Linear; Slope = -46.34, 95% CI 2-sided [-88.5 to -4.18]
Statistical Analysis 13: Comparison: Exposure-based Therapy vs Behavioral Activation Therapy; Change in conflict arbitration response time (AAC conflict RT post-pre) predicting trajectories of PSWQ scores over the 10 sessions: RT_change main effect; Test type: Other; p = .546, Regression, Linear; Slope = 39.53, 95% CI 2-sided [-94.2 to 173.85]
Statistical Analysis 14: Comparison: Exposure-based Therapy vs Behavioral Activation Therapy; Change in conflict arbitration response time (AAC conflict RT post-pre) predicting trajectories of PSWQ scores over the 10 sessions: Treatment x RT_change interaction; Test type: Superiority; p = .443, Regression, Linear; Slope = -89.96, 95% CI 2-sided [-327.39 to 147.67]

7. Secondary Outcome: Depressive Symptoms as Measured by the Beck Depression Inventory - II.
Description: Test the predictive effects of imaging and behavioral factors on symptoms at post-treatment (within 6 weeks after completing treatment), covarying for baseline symptom severity. The BDI-II is a 21-item questionnaire, with each individual item being rated from 0-3 in a list of four statements arranged in increasing severity about a particular symptom of depression. The outcome measure is the total score on the BDI-II, which is the sum of all 21 items. Higher scores equate to greater severity of depression symptoms. Total score of 0-13 is considered minimal range, 14-19 is mild, 20-28 is moderate, and 29-63 is severe.
Time Frame: as for outcome 6
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Exposure-based Therapy | Behavioral Activation Therapy
Number analyzed (Participants) | 27 | 29
score on a scale | 13.56 (6.95) | 9.68 (8.64)
Statistical Analysis 1: Comparison: Exposure-based Therapy vs Behavioral Activation Therapy; Relationships between baseline average approach behavior during conflict trials on the AAC and post-treatment BDI-II score: approach behavior main effect; Test type: Other; p = .357, Regression, Linear; Slope = -1.01, 95% CI 2-sided [-3.22 to 1.19]
Statistical Analysis 2: Comparison: Exposure-based Therapy vs Behavioral Activation Therapy; Relationships between baseline average approach behavior during conflict trials on the AAC and post-treatment BDI-II score: treatment x approach behavior interaction; Test type: Superiority; p = .812, Regression, Linear; Slope = .37, 95% CI 2-sided [-2.74 to 3.47]
Statistical Analysis 3: Comparison: Exposure-based Therapy vs Behavioral Activation Therapy; Relationships between baseline average RT during conflict trials on the AAC and post-treatment BDI-II score: RT main effect; Test type: Other; p = .826, Regression, Linear; Slope = 2.01, 95% CI 2-sided [-16.42 to 20.45]
Statistical Analysis 4: Comparison: Exposure-based Therapy vs Behavioral Activation Therapy; Relationships between baseline average RT during conflict trials on the AAC and post-treatment BDI-II score: treatment x RT interaction; Test type: Superiority; p = .838, Regression, Linear; Slope = -2.89, 95% CI 2-sided [-31.42 to 25.64]
Statistical Analysis 5: Comparison: Exposure-based Therapy vs Behavioral Activation Therapy; Relationship of striatum activity during points outcomes (reward) with BDI-II post-treatment: striatum main effect; Test type: Other; p = .776, Regression, Linear; Slope = -0.68, 95% CI 2-sided [-5.51 to 4.14]
Statistical Analysis 6: Comparison: Exposure-based Therapy vs Behavioral Activation Therapy; Relationship of striatum activity during points outcomes (reward) with BDI-II post-treatment: treatment x striatum interaction effects; Test type: Superiority; p = .844, Regression, Linear; Slope = -0.69, 95% CI 2-sided [-7.79 to 6.40]
Statistical Analysis 7: Comparison: Exposure-based Therapy vs Behavioral Activation Therapy; Relationship of right amygdala activity during negative images with BDI-II post-treatment: amygdala main effect; Test type: Other; p = .719, Regression, Linear; Slope = .88, 95% CI 2-sided [-4.03 to 5.79]
Statistical Analysis 8: Comparison: Exposure-based Therapy vs Behavioral Activation Therapy; Relationship of right amygdala activity during negative images with BDI-II post-treatment: treatment x amygdala interaction; Test type: Superiority; p = .464, Regression, Linear; Slope = -2.33, 95% CI 2-sided [-8.74 to 4.07]
Statistical Analysis 9: Comparison: Exposure-based Therapy vs Behavioral Activation Therapy; Relationship of right dlPFC activity during negative images with BDI-II post-treatment: dlPFC main effect; Test type: Other; p = .135, Regression, Linear; Slope = 5.91, 95% CI 2-sided [-1.93 to 13.75]
Statistical Analysis 10: Comparison: Exposure-based Therapy vs Behavioral Activation Therapy; Relationship of right dlPFC activity during negative images with BDI-II post-treatment: treatment x dlPFC interaction; Test type: Superiority; p = .158, Regression, Linear; Slope = -6.09, 95% CI 2-sided [-14.65 to 2.47]
Statistical Analysis 11: Comparison: Exposure-based Therapy vs Behavioral Activation Therapy; Change in behavior (AAC conflict post-pre) predicting trajectories of BDI-II cores over the 10 sessions: Behavior_change main effect; Test type: Other; p = .690, Regression, Linear; Slope = 1.16, 95% CI 2-sided [-4.78 to 7.11]
Statistical Analysis 12: Comparison: Exposure-based Therapy vs Behavioral Activation Therapy; Change in behavior (AAC conflict post-pre) predicting trajectories of BDI-II scores over the 10 sessions: Treatment x Behavior_change interaction; Test type: Superiority; p = .715, Regression, Linear; Slope = -1.37, 95% CI 2-sided [-8.99 to 6.25]
Statistical Analysis 13: Comparison: Exposure-based Therapy vs Behavioral Activation Therapy; Change in conflict arbitration response time (AAC conflict RT post-pre) predicting trajectories of BDI-II scores over the 10 sessions: RT_change main effect; Test type: Other; p = .740, Regression, Linear; Slope = 5.14, 95% CI 2-sided [-26.38 to 36.65]
Statistical Analysis 14: Comparison: Exposure-based Therapy vs Behavioral Activation Therapy; Change in conflict arbitration response time (AAC conflict RT post-pre) predicting trajectories of BDI-II scores over the 10 sessions: Treatment x RT_change interaction; Test type: Superiority; p = .966, Regression, Linear; Slope = -0.98, 95% CI 2-sided [-48.10 to 46.14]

ADVERSE EVENTS:
Time Frame: From pre- to post-treatment: post-treatment timepoint assessed within 6 weeks following last treatment session, on average 16 weeks after baseline assessment
Groups:
- Exposure-based Therapy: Participants will complete 10, 90-minute sessions of Exposure-based therapy, conducted using a group format. Each group will include 8-12 participants. Exposure-based therapy seeks to increase abilities to manage anxiety through repeated practice in facing the situations or thoughts that are the focus of worry or fear. All participants will complete computer-based behavioral assessments, surveys and interviews, functional magnetic resonance imaging (fMRI), and electroencephalography (EEG).
  Exposure-based therapy: Exposure-based therapy
  Computer-based behavioral assessment: Computer-based tasks during which participants respond to images on the screen, including abstract images, emotional faces, and pleasant and unpleasant images.
  Surveys and Interviews: Surveys and interviews in which participants will be asked to answer questions related to their mental and physical health history and current symptoms.
  Magnetic resonance imaging (MRI): Magnetic resonance imaging (MRI) will be used to obtain information concerning the structure of the brain, as well as to assess changes associated with blood flow in the brain while participants are completing behavioral tasks (see description of computer-based behavioral assessment intervention).
  Electroencephalography (EEG): Electroencephalography (EEG) will be used to assess changes in electrical activity of the brain while participants complete behavioral tasks (see description of computer-based behavioral assessment).
Arm/Group | Exposure-based Therapy | Behavioral Activation Therapy
All-Cause Mortality (participants affected / at risk) | 0/46 | 0/48
Serious Adverse Events (participants affected / at risk) | 0/46 | 0/48
Other Adverse Events (participants affected / at risk) | 0/46 | 1/48
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Exposure-based Therapy (N=46) | Behavioral Activation Therapy (N=48)
Active suicidal ideation (Psychiatric disorders) | 0 (0) | 1 (1) — One participant in BA reported active suicidal ideation at one treatment timepoint (endorsing "I would like to kill myself" on the BDI-II suicidal ideation item). Risk assessment determined participant was safe to continue in the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-03-13): https://cdn.clinicaltrials.gov/large-docs/80/NCT02807480/Prot_000.pdf
  • Informed Consent Form (2019-06-24): https://cdn.clinicaltrials.gov/large-docs/80/NCT02807480/ICF_001.pdf